CLINICAL TRIAL: NCT01112280
Title: Prospective Randomized Controlled Trial of Cap-Assisted ChromoEndoscopy(CapACE) Versus Conventional Colonoscopy(CC) for the Detection of Colorectal Neoplasia
Brief Title: Efficacy of Cap-assisted Chromoendoscopy as a Screening Test for Colorectal Neoplasm Using Web-based Research Network
Acronym: CapACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korean Association for the Study of Intestinal Diseases (Other)
Collaborators: National Cancer Center, Korea (Other Government); Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Hyun-Soo Kim, Professor, Korean Association for the Study of Intestinal Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KASID polyp-01; MHWFA A092230 (Other Grant/Funding Number: Ministry of Health, Welfare & Family Affairs, Korea)
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Neoplasm
Keywords: Colorectal neoplasm; Colonoscopy; chromoendoscopy; cap-assisted colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cap-assisted chromoendoscopy (Experimental): To the tip of the colonoscope, transparent cap is fitted and applied. In addition, panchromoendoscopy using indigocarmine solution is preformed in this group.
  Interventions: Device: cap-assisted chromoendoscopy
- Standard colonoscopy (No Intervention): Neither transparent cap nor chromoendoscopy is applied in this group and standard colonoscopy is performed.

INTERVENTIONS:
Device: cap-assisted chromoendoscopy — A cap (irrigation cap) is a simple plastic device that can be attached to the tip of a colonoscope before performing the colonoscopy. For chromoendoscopy, 0.09% indigocarmine was administered via irrigation cap .
  Arms: cap-assisted chromoendoscopy

SUMMARY:
The investigators plan to conduct a multi-center, randomized controlled trial to investigate the efficacy of cap-assisted chromoendoscopy as a screening test for detection of colorectal polyp. This study will be performed using web-based research network, e-VELOS in Korea.

DETAILED DESCRIPTION:
Various endoscopic tools have been tried to reduce polyp missing rate which has been reported to be 20-25%. Transparent cap-assisted colonoscopy has been suggested to improve visualization of the lesion that are difficult to access, such as tangentially located lesions and those located within a limited luminal space. Chromoendoscopy with indigocarmine spraying was reported to increases the detection rates of polyp, especially in right colon and rectum. However, there also have been mixed results regarding polyp detection rates of the endoscopic methods. Moreover, there is no data regarding the impact of the screening tools on longterm recurrence rate of colorectal polyp. Therefore, in this study, we intend to perform a multi-center, randomized controlled trial to investigate the efficacy of cap-assisted chromoendoscopy as a screening test for detection of colorectal polyps. This study will be performed using web-based research network, e-VELOS in Korea.

ELIGIBILITY:
Inclusion Criteria:

* All asymptomatic colonoscopic examinees

Exclusion Criteria:

* Familial history of hereditary colorectal cancer
* History of colorectal cancer
* Patients had received colonoscopy examination before
* Familial or past history of FAP(familiar adenomatous polyposis)
* Colonic polyposis syndrome
* Prior colonic resection of any part of the colon
* Allergy to indigo carmine
* Inflammatory bowel disease
* Pregnancy
* Inability to provide informed consent

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1905 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 7 days is needed to confirm the pathologic examination.
  The proportion of subjects with at least one adenoma

SECONDARY OUTCOMES:
Proximal adenoma detection rate | 7 days is needed to confirm the pathologic examination.
  Proportion of subjects with at least one proximal colon adenoma
Proximal serrated polyp detection rate | 7 days is needed to confirm the pathologic examination.
  Proportion of subjects with at least one proximal serrated polyp/adenoma
Advanced adenoma detection rate | 7 days is needed to confirm the pathologic examination.
  Proportion of subjects with at least one advanced adenoma
Serrated adenoma detection rate | 7 days is needed to confirm the pathologic examination.
  Proportion of subjects with at least one serrated adenoma
Cancer detection rate | 7 days is needed to confirm the pathologic examination.
  Proportion of subjects with at least one cancer
Surveillance | 7 - 14 days
  Surveillance interval recommendations for both groups were classified based on adenoma detection

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Soo Kim, Principal Investigator — Korean Association for the Study of Intestinal Diseases
Locations (14):
- South Korea (14):
  - Hallym University Medical Center, Anyang
  - Kosin University College of Medicine, Busan
  - Dankuk University college of medicine hospital, Cheonan
  - National Cancer Center Hospital, National Cancer Center, Goyang
  - Hanyang University Guri Hospital, Hanyang University College of Medicine, Guri-si
  - Catholic university St. Mari's hospital, Incheon
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul
  - Ewha Mokdong hospital, Seoul
  - Kyung Hee University Hospital at Gang Dong, Kyung Hee University School of Medicine, Seoul
  - Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul
  - Sunchunhyang University hospital, Seoul
  - Sungkyunkwan University Kangbuk Samsung hospital, Seoul
  - Yonsei University College of Medicine, Seoul
  - Yonsei Uiniversity Wonju College of Medicine, Wŏnju

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim SY, Park HJ, Kim HS, Park DI, Cha JM, Park SJ, Choi H, Shin JE, Eun CS, Kim JO, Kim HG, Kim SE, Park CH, Kim TI, Hong SN. Cap-Assisted Chromoendoscopy Using a Mounted Cap Versus Standard Colonoscopy for Adenoma Detection. Am J Gastroenterol. 2020 Mar;115(3):465-472. doi: 10.14309/ajg.0000000000000510. PMID 31972618